CLINICAL TRIAL: NCT04657978
Title: High Density Substrate Evaluation and Guided Ablation Therapy for Atrial Fibrillation
Brief Title: Substrate Guided Ablation Therapy for Atrial Fibrillation
Acronym: HEAT-AF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 263083
Record Dates: First submitted 2020-11-27; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Atrial fibrillation; Catheter Ablation; Substrate
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Substrate guided intervention arm: Participants recruited to the study will undergo High Density Wave Solution™ guided substrate mapping of the left atrium. Ablation will thereafter be performed to comprise wide area circumferential ablation of the pulmonary veins in pairs, followed by ablation of low voltage zones in the left atrium.
  Interventions: Procedure: Substrate guided left atrial ablation

INTERVENTIONS:
Procedure: Substrate guided left atrial ablation — Ablation therapy targeting areas of low voltage, which may include encirclement, homogenization or targeting of abnormal electrograms and anchored to a non-conducting structure if the region is in close proximity or likely to create an isthmus for arrhythmias.

SUMMARY:
Atrial fibrillation (AF), often referred to as an 'irregular heartbeat', is the most common abnormal heart rhythm worldwide. AF may be intermittent (termed paroxysmal) or sustained (termed persistent).Catheter ablation is increasingly being used to manage individuals with AF, however in a significant proportion of cases AF recurs. Such rhythm control interventions are known to be less effective in individuals with persistent AF compared with those with paroxysmal AF. Analysis of heart tissue of individuals with AF show deposition of scar tissue within the heart muscle and this scar tissue promotes abnormal electrical activity that is involved in causing AF. The aim of the proposed study is to evaluate the feasibility and effectiveness of combining conventional pulmonary vein isolation (PVI) during catheter ablation for AF with adjunctive substrate ablation.

DETAILED DESCRIPTION:
This is a single-centre, non-randomized study investigating the feasibility, safety and efficacy of substrate guided ablation in persistent AF.

The study population will be patients between the ages of 18 and 80 with symptomatic, persistent atrial fibrillation (≥1 year) referred for catheter ablation on standard clinical grounds.

The catheter ablation procedure will be performed using the Precision Ensite™ three dimensional mapping system and the Advisor High Density Grid™ mapping catheter (Abbott Medical Incorporated). All patients will undergo conventional pulmonary vein isolation (PVI). As an adjunctive strategy to PVI, low voltage areas (used as a surrogate for atrial scar), as derived from the voltage map, will be targeted for ablation in order to isolate or homogenise these areas of the atrium. A pre-procedural cardiac magnetic resonance imaging scan will be performed in all patients.

All patients will undergo 12 months follow-up with an ECG and ambulatory holter monitoring at 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years and ≤ 80 with a clinical indication for persistent atrial fibrillation ablation

Exclusion Criteria:

* Contraindication to anticoagulation
* Thrombus in the left atrium despite anticoagulation
* Cerebrovascular accident within the previous 6 months
* Patients actively participating in another research study will be not be permitted to enrol. Patients who have been involved with other research studies will be able to participate after a minimum period of 3 months after completion of prior study follow up
* Females of childbearing potential must have a negative pregnancy test on the day of the ablation procedure due to the radiation exposure during the procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from patients with persistent atrial fibrillation who have been referred for catheter ablation based on standard clinical grounds.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial arrhythmias (>30 seconds) after a single procedure without anti-arrhythmic drugs (AADs) within 12 months, measured by ambulatory holter monitoring | 12 month
  All participants will have an ECG and ambulatory holter monitor performed at 3, 6 and 12 months after the procedure.

SECONDARY OUTCOMES:
To compare 1-year arrhythmia free clinical outcome with historical control patients matched by propensity score | 12 Months
  Freedom from AF defined as no documented AF (>30 seconds) following the 3 months blanking period following a single procedure, off anti-arrhythmic drugs.
Safety endpoint evaluating the incidence of intraprocedural (primarily Advisor High Density Grid™ mapping catheter) related adverse events | 12 Months
To correlate cardiac MRI derived scar distribution and burden in the left atrium with the baseline voltage map obtained using the Advisor High Density Grid™ catheter | 12 Months
  The left atrium will be segregated into pre-defined regions and marked for presence or absence of fibrosis as identified on MRI scans and low voltage identified on invasive mapping. Inter-class correlation will performed to evaluate consistency between modalities.

CONTACTS AND LOCATIONS:
Overall Officials: Shouvik Haldar, FRCP MD, Principal Investigator — Royal Brompton and Harefield Hospital

IPD SHARING:
Plan to Share IPD: No